CLINICAL TRIAL: NCT02180334
Title: The Effect of Combination of Mosapride and Dipeptidyl Peptidase-4 (DPP-4) Inhibitor on Plasma Concentration of Incretin Hormones
Brief Title: The Effect of Combination of Mosapride and DPP-4 Inhibitor on Plasma Concentration of Incretin Hormones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-1311-104-537; 2013-2641 (Other: SNUH Institutional Review Board)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2014-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Gastric Emptying; Gastrointestinal Motility; Incretins; Glucagon-Like Peptide 1; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — mosapride; Linagliptin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mosapride (Experimental): * Mosapride citrate 5 mg (Gasmotin®): 1 tablet (5 mg) will be administered 1 hour before MMTT.
  * Linagliptin 5 mg (Trajenta®): 1 tablet (5 mg) per day should be taken for 7 days during run-in period. 1 tablet (5 mg) will be administered 1 hour before MMTT.
  * Acetaminophen 500 mg (Tylenol®): 3 tablets (1500 mg) will be administered at once with the mixed meal for calculating gastric emptying time.
  Interventions: Drug: Mosapride citrate; Drug: Linagliptin; Drug: Acetaminophen (paracetamol)
- Control (Placebo Comparator): * Placebo drug: 1 tablet will be administered 1 hour before MMTT.
  * Linagliptin 5 mg (Trajenta®): 1 tablet (5 mg) per day should be taken for 7 days during run-in period. 1 tablet (5 mg) will be administered 1 hour before MMTT.
  * Acetaminophen 500 mg (Tylenol®): 3 tablets (1500 mg) will be administered at once with the mixed meal for calculating gastric emptying time.
  Interventions: Drug: Linagliptin; Drug: Acetaminophen (paracetamol)

INTERVENTIONS:
Drug: Mosapride citrate — On the day of MMTT, 1 tablet (5 mg) of mosapride will be administered orally to participants of 'mosapride' arm. After 1 hour, MMTT will be performed.
  Other Names: Gasmotin®
  Arms: Mosapride
Drug: Linagliptin — During run-in period, 1 tablet (5mg) per day will provided for 7 days. On the day of MMTT, 1 tablet (5 mg) of linagliptin will be administered orally to participants of both arms. After 1 hour, MMTT will be performed.
  Other Names: Trajenta®
Drug: Acetaminophen (paracetamol) — On the day of MMTT, 3 tablets (1500 mg) of acetaminophen (paracetamol) will be administered orally to participants of both arms at the start of MMTT with manufactured mixed meal (0 min).
  Other Names: Tylenol®

SUMMARY:
The aim of this study is to investigate the effects of combined administration of mosapride as modulator of gastrointestinal motility and DPP-4 inhibitor on secretion of gut hormone such as glucagon-like peptide-1 (GLP-1) and gastric inhibitory polypeptide (GIP), and oral glucose tolerance. Additionally, change in lipid profile and insulin secretion will be also assessed.

DETAILED DESCRIPTION:
This is randomized, double-blind, placebo-controlled, cross-over study. After screening and enrollment, participants will take 5 mg of linagliptin once a day for one week of run-in period (Day 1 to Day 7). Randomization will be done on Day 8 to assign the participants to either mosapride arm or placebo arm. If a subject is assigned to mosapride arm, mixed meal tolerance test (MMTT) will be performed after taking mosapride with linagliptin. If a subject is assigned to placebo arm, he/she will take placebo instead of mosapride before MMTT. On Day 9, all subjects will be crossed over to the other arm and MMTT will proceed with medication depending on their arms. Gastric emptying time measurement with paracetamol will be done along with MMTT. Plasma incretin hormone levels in two arms will be compared.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* BMI < 35 kg/m2
* HbA1c 6.5~8.0% for whom is on lifestyle modification only, 6.0~8.0% for whom is taking oral antidiabetic drug(s).
* on lifestyle modification or oral antidiabetic therapy (sulfonylurea, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, and DPP-4 inhibitors)
* Who read and signed the informed consent agreement

Exclusion Criteria:

* chronic disease(s) requiring medication other than diabetes mellitus
* type 1 diabetes mellitus or history of diabetic ketoacidosis
* on insulin therapy or requiring insulin therapy
* history of gastrointestinal surgery excluding appendectomy, hernia repair and hemorrhoid surgery
* serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) to be more than 2.5 times above the upper limit of normal
* estimated glomerular filtration rate to be less than 50 mL/min/1.73m2
* genetic disorders associated with digestion and absorption such as galactose intolerance, Lapp lactase deficiency, and glucose-galactose malabsorption
* history of hypersensitivity including anaphylaxis and angioedema to mosapride citrate, linagliptin, or paracetamol (acetaminophen)
* history of asthma associated with aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)
* currently taking drugs that can prolong QT interval, including procainamide, quinidine, flecainide, sotalol, tricyclic antidepressants
* currently taking anticholinergics such as atropine sulfate, scopolamine butylbromide
* child-bearing or lactating women
* women in reproductive age who disagree with contraception with proper method or urine pregnancy test during the study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of plasma total GLP-1 levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma total GLP-1 levels during MMTT

SECONDARY OUTCOMES:
Area under the curve (AUC) of plasma total GIP levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma total GIP levels during MMTT
Area under the curve (AUC) of plasma glucose levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma glucose levels during MMTT
Area under the curve (AUC) of plasma insulin levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma insulin levels during MMTT
Area under the curve (AUC) of plasma C-peptide levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma C-peptide levels during MMTT
Area under the curve (AUC) of serum triglyceride levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of serum triglyceride levels during MMTT
Area under the curve (AUC) of serum nonesterified fatty acid (NEFA) levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of serum NEFA levels during MMTT
Area under the curve (AUC) of plasma active GLP-1 levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma active GLP-1 levels during MMTT

OTHER OUTCOMES:
Area under the curve (AUC) of plasma paracetamol levels | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  AUC of plasma paracetamol levels during MMTT
The peak concentration of plasma paracetamol | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  The peak concentration of plasma paracetamol during MMTT
The time to peak concentration of plasma paracetamol | 0, 15, 30, 60, 90, 120, 150, 180 min after taking mixed meal (manufactured)
  The time to peak concentration of plasma paracetamol during MMTT

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Study Chair — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea